CLINICAL TRIAL: NCT01863238
Title: An Ocular Safety Study of Ivacaftor-Treated Pediatric Patients 11 Years of Age or Younger With Cystic Fibrosis
Status: Completed | Type: Observational
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: VX12-770-115
Record Dates: First submitted 2013-05-22; First posted 2013-05-27 (Estimated); Last update posted 2016-08-23 (Estimated); Status verified 2015-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Ivacaftor Treated
  Interventions: Other: Ophthalmologic examinations; Drug: Ivacaftor Exposed

INTERVENTIONS:
Other: Ophthalmologic examinations — Subjects will undergo an ophthalmologic examination at study entry (Day 1) and every 6 months thereafter for 2 years (Months 6, 12, 18, and 24). Subjects who discontinue treatment with commercially-available ivacaftor for any reason and are willing to continue participation in the study will complete the study.
Drug: Ivacaftor Exposed

SUMMARY:
This study is designed to evaluate the risk of cataracts (lens opacities) and describe the best corrected distance vision (with glasses/contacts for those who wear them) of pediatric patients with Cystic Fibrosis who are 11 years of age or younger at the time of ivacaftor treatment initiation and are receiving or planning to receive commercially-available ivacaftor in the US.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 11 years of age or younger at the time of treatment initiation with ivacaftor (as part of clinical trial) or commercially-available ivacaftor.
2. Subject must reside in the US and be receiving or planning to receive commercially-available ivacaftor.

Exclusion Criteria:

1. Subject is enrolled in an ivacaftor clinical study in which ivacaftor exposure is mandated by the protocol.
2. Subject has received surgery for cataracts

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patients with CF who are 11 years of age or younger at the time of initiation of treatment with ivacaftor and are receiving or planning to receive commercially-available ivacaftor in the United States (US)
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2013-05; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Cataracts (lens opacities) | Through Month 24
Best corrected distance vision | Through Month 24

CONTACTS AND LOCATIONS:
Locations (38):
- United States (38):
  - Birmingham, Alabama
  - Tucson, Arizona
  - Long Beach, California
  - Aurora, Colorado
  - Wilmington, Delaware
  - St. Petersburg, Florida
  - Boise, Idaho
  - Chicago, Illinois
  - Indianapolis, Indiana
  - Kansas City, Kansas
  - Louisville, Kentucky
  - Portland, Maine
  - Boston, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Columbia, Missouri
  - Kansas City, Missouri
  - Omaha, Nebraska
  - Rochester, New York
  - Akron, Ohio
  - Cincinnati, Ohio
  - Toledo, Ohio
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Providence, Rhode Island
  - Charleston, South Carolina
  - Knoxville, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Charlottesville, Virginia
  - Seattle, Washington
  - Spokane, Washington
  - Morgantown, West Virginia